CLINICAL TRIAL: NCT04420416
Title: dePression, Anxiety, aNd acaDemic pErforMance In Covid-19: PANDEMIC Study.
Brief Title: Mental Health and Academic Performance in COVID-19
Acronym: PANDEMIC
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Investigador Titular D, Instituto Mexicano del Seguro Social
Other Study IDs: Mental01
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Depression, Anxiety
Keywords: COVID-19; Depression; Anxiety; Public health; Academic performance
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — The investigators will use the Spanish language validated version of the Academic Self-Concept Scale (ASCS), the Patient Health Questionnaire-9 (PHQ-9) depression screening scale, and the General Anxiety Disorder-7 (GAD-7) screening scale. Additionally, the sample will be asked about their gender, age, preference of teaching modality, and finally, if the participants have perceived a change in their performance or any change in their grades.

SUMMARY:
This study aims to identify the preference of the class modalities (classroom or online) in undergraduate and graduate students. Additionally, to explore if the presence of any mental state alterations such as depression or anxiety due to the COVID-19 pandemic can alter their perception of academic performance.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Students of any undergraduate or graduate course who are attending their semester online

Exclusion Criteria:

* Students who are not attending an online course
* Students who are not registered in a university undergraduate or graduate course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Undergraduate and graduate students who attend an online university course.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Academic Self-Concept Scale Score | up to 3 months
  This scale will explore the effort and confidence of the participants. The minimum score for each facet is 10, and the maximum score is 70.
PHQ-9 Score | up to 3 months
  This inventory will be used to identify the presence and intensity of depressive disorders. The minimum score is 0, and the maximum score is 27.
GAD-7 Score | up to 3 months
  This questionnaire will be used to evaluate the presence and intensity of anxiety disorders. The minimum score is 0, and the maximum score is 21.
Preference of teaching method | up to 3 months
  Students' preference of classroom or online classes.
Self perceived academic performance | up to 3 months
  Students' perception of changes in their academic performance: got better, worse, or stayed the same.
Academic grades changes | up to 3 months
  Students' perception of changes in their grades: got better, worse, or stayed the same.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no plan of making individual participant data available.